CLINICAL TRIAL: NCT07040150
Title: Development and Short-Term Evaluation of a Novel Semi-Rigid Brace for Adolescent Idiopathic Scoliosis: Results From a Multicenter Prospective Observational Study of the First 60 Patients
Brief Title: Evaluation of a Novel Semi-Rigid Brace for Adolescent Idiopathic Scoliosis
Status: Active, not recruiting | Type: Observational
Sponsor: Nippon Sigmax co., ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: AMEC brace study
Record Dates: First submitted 2025-06-25; First posted 2025-06-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Spinal bracing — The semi-rigid spinal brace was developed to enhance patient compliance while maintaining effective curve correction. Patients were instructed to wear the brace for 18-20 h daily.

SUMMARY:
Introduction: Spinal bracing remains the gold standard for conservative management of adolescent idiopathic scoliosis (AIS). However, poor adherence often limits treatment efficacy. The development of a brace that enhances compliance while maintaining sufficient corrective force is crucial. This study aimed to develop and evaluate the effectiveness of a novel semi-rigid brace for AIS based on wearing time and correction rate.

Materials and Methods: The investigators enrolled patients who met the following Scoliosis Research Society (SRS) criteria for brace treatment: (1) confirmed AIS diagnosis, (2) Risser sign ≤ 2, (3) Cobb angle between 25° and 40°, (4) age ≥ 10 years, and (5) single-curve pattern. Wearing time was objectively measured over 180 days using embedded temperature sensors. Correction rates were assessed at initiation and after 180 days or more.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed AIS
* Risser sign ≤ 2
* Cobb angle between 25° and 40°
* age ≥ 10 years
* single-curve pattern (thoracic or thoracolumbar/ lumbar)
* premenarchial or less than one year post-menarche.

Exclusion Criteria:

* Patients who do not meet the SRS criteria for orthosis suitability
* Patients with a history of spinal surgery

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Conducted at seven medical institutions in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Wearing time | 180 days from registration

SECONDARY OUTCOMES:
Initial correction rate | Immediately after registration
Correction rate after 180 days or more | 180 days or more from registration
Treatment success rate | 2 years or more from registration

CONTACTS AND LOCATIONS:
Locations (1):
- Aizu Medical Center at Fukushima Medical University, Aizu-Wakamatsu, Fukushima, Japan

IPD SHARING:
Plan to Share IPD: No
The investigators will not be sharing individual participant data (IPD) due to privacy concerns.

REFERENCES:
- [Background] Richards BS, Bernstein RM, D'Amato CR, Thompson GH. Standardization of criteria for adolescent idiopathic scoliosis brace studies: SRS Committee on Bracing and Nonoperative Management. Spine (Phila Pa 1976). 2005 Sep 15;30(18):2068-75; discussion 2076-7. doi: 10.1097/01.brs.0000178819.90239.d0. PMID 16166897
- [Background] Struhl K, Chen W, Hill DE, Hope IA, Oettinger MA. Constitutive and coordinately regulated transcription of yeast genes: promoter elements, positive and negative regulatory sites, and DNA binding proteins. Cold Spring Harb Symp Quant Biol. 1985;50:489-503. doi: 10.1101/sqb.1985.050.01.061. No abstract available. PMID 3913566